CLINICAL TRIAL: NCT04457531
Title: A Randomized Controlled Study of LiuWeiLuoBi Granule for the Treatment of Diabetic Peripheral Neuropathy
Brief Title: LiuWeiLuoBi Granule for the Treatment of Diabetic Peripheral Neuropathy
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Zhong Wang, Professor, China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LIUWEI-V1.1
Record Dates: First submitted 2020-03-15; First posted 2020-07-07 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Diabetic Peripheral Neuropathy; Chinese Medicine; Nerve Conduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LiuWeiLuoBi Group (Experimental): Patients will receive the treatment of LiuWeiLuoBi Granule for 12 weeks,twice a day added to the standard medical treatment.
  Interventions: Drug: LiuWeiLuoBi Granule; Other: Standard medical treatment
- Control Group (Other): Patients will receive the standard medical treatment for 12 weeks.
  Interventions: Other: Standard medical treatment

INTERVENTIONS:
Drug: LiuWeiLuoBi Granule — LiuWeiLuoBi Granule is a Chinese medicine made from 6 herbal medicine, including Shaji(Sea-buckthorn), Honghua (Safflower), Jinyinhua(Honeysuckle),etc.
  Arms: LiuWeiLuoBi Group
Other: Standard medical treatment — Standard medical therapy is adhered to the guidline issued by American Diabetes Association and Chinese Diabetes Society at 2017, including keeping an appropriate diet, doing some exercises, the pharmacological therapy to control the blood glucose, blood pressure and blood lipids.

SUMMARY:
Based on network pharmacology, Liuweiluobi Granule was screened to treat diabetes peripheral neuropathy with deficiency of the spleen and kidney and stasis-heat syndrome.In the preliminary animal experiment, it suggested that this granule had a significant protective effect on the peripheral motor nerves of diabetic peripheral neuropathy and the effect of anti-inflammation, and the prescription did not induce the death of zebrafish at a concentration of 1000 ug/mL, without any obvious toxicity. This study aims to evaluate the efficacy of Liuweiluobi Granule in improving neurotransmission function in patients with diabetic peripheral neuropathy through a pilot, randomized controlled study.

ELIGIBILITY:
Inclusion criteria

1. Meet the clinical confirmed diagnostic criteria of "diabetic peripheral neuropathy";
2. Toronto score ≥ 6 points;
3. Meet the Chinese medicine diagnostic criteria of Pi-Shen-Liang-Xu (Deficiency of Pi and Shen) and Yu-Re-Ru-Luo (Collaterals with Stasis and Heat） Zheng (Syndrome) in diabetic peripheral neuropathy;
4. Over 18 years old and under 75 years old, regardless of gender and ethnicity;
5. Have received basic treatment for diabetes controled with stable blood glucose level (fasting blood glucose: <7mmol / L; 2h postprandial blood glucose: <11.1mmol / L; glycated hemoglobin: <8%);
6. Have not taken or stopped taking DPN-related drugs (Mutan granules, Qidan Tongluo granules, pregabalin, duloxetine, etc.) for more than one week;
7. Sign the informed consent form with valid telephone contact information.

Exclusion criteria

1. Patients with diabetic ketosis, ketoacidosis or co-infection;
2. Patients with known malignant tumors;
3. Patients with known severe brain diseases, as cerebral infactions with limited activity；
4. Patients with known severe arrhythmias or heart failure over Grade 2 (New York Heart Association), or other known severe heart diseases;
5. Patients with known severe kidney impairment (creatinine ≥200ummol/L);
6. During the screening or within 24 hours before screening, patients were found to have any of the following laboratory parameter abnormalities (based on local laboratory reference range):-ALT and/or AST level> 2 times the upper limit of normal range (ULN);
7. Patients with spinal cord injury, cervical and lumbar spine lesions (nervous root compression, spinal stenosis, cervical and lumbar degenerative lesions) or sequelae of cerebrovascular disease, neuromuscular junction or muscle disease;
8. Patients with other neuropathy diseases caused by, such as: cerebral infarction, Guillain-Barre syndrome, severe arteriovenous vascular disease (venous embolism, lymphangitis), chronic inflammatory demyelinating polyneuropathy, VitB Deficiency, hypothyroidism, alcoholism, neurotoxicity indused by chemotherapeutic drugs, or metabolic nerve damage caused by renal insufficiency;
9. Patients with severe arteriovenous vascular disease (venous embolism, lymphangitis, etc.);
10. Patients with epilepsy or mental illness;
11. Alcoholics;
12. Patients with a history of psychotropic substance abuse;
13. Patients with allergies or allergies to any drugs in the trial;
14. pregnant women or patients with intention to become pregnant;
15. Participated in other clinical trials in the past 1 month;
16. Patients would not take drug continuously which could affect the evaluation of efficacy;
17. Investigator evaluates as unsuitable to participate in this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-10-26 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Mean maximal nerve conduction velocity | 12 weeks
  Mean maximal conduction velocity of the common peroneal motor nerve (MCV) and sensory nerve (SCV)

SECONDARY OUTCOMES:
Michigan Diabetic Peripheral Neuropathy Score (MDNS) | Baseline, 4 weeks, 8 weeks and 12 weeks
  Michigan Diabetic Peripheral Neuropathy Score (MDNS) is a 46 point clinical score, with score ranging from 0 to 3 (score of 0, normal; 1, mild to moderate; 2, severe and score of 3, absent). The score is more high means a worse outcome.In MDNS vibration, pain, and light touch are assessed with a 128 Hz tuning fork, a pin, and a 10g filament, respectively. The outcome measures were performed by the investigator at baseline and at the eighth week.
Toronto clinical scoring system (TCSS) | Baseline, 4 weeks, 8 weeks and 12 weeks
  Toronto clinical scoring system (TCSS) includes three parts: the symptom score of the symptom, the reflection score of the nerve and the evaluation score of the sensory function test. Symptoms include numbness, pain, and needle-like sensation in the lower extremities Feelings of weakness, weakness, instability in walking, and similar symptoms of the upper limbs, such as normal score of 0, 1 point for the presence of corresponding symptoms, a total of 6 points; nerve reflex including ankle reflex and knee reflex, bilateral score, normal score of 0, weakened 1 point, 2 points for disappearance, 8 points in total; sensory function test includes 5 items of pain, temperature, pressure, vibration, and position on the right big toe, 0 points for normal, 1 point for abnormality, 5 points in total With a total score of 19 points. With a score of 0 to 5 do not exist in the DPN, 6 to 8 are mild DPN, 9 to 11 are moderate DPN, 12 to 19 are severe DPN.
Quantitative symptoms scales of DPN in Traditional Chinese medicine | Baseline, 4 weeks, 8 weeks and 12 weeks
HbA1c | Baseline, 4 weeks, 8 weeks and 12 weeks
Changes in the level of aldose reductase | to 12 weeks
Fasting blood glucose | Baseline, 4 weeks, 8 weeks and 12 weeks
2 hrs postprandial blood glucose | Baseline, 4 weeks, 8 weeks and 12 weeks
Total lipids (TC) | Baseline, 4 weeks, 8 weeks and 12 weeks
  Lipid level
triglycerides (TG) | Baseline, 4 weeks, 8 weeks and 12 weeks
  Lipid level
high density lipoprotein cholesterol (HDL-C) | Baseline, 4 weeks, 8 weeks and 12 weeks
  Lipid level
low density lipid Protein cholesterol (LDL-C). | Baseline, 4 weeks, 8 weeks and 12 weeks
  Lipid level

OTHER OUTCOMES:
Amino acids, lipid metabolites, vitamins, neurotransmitters and other metabolites | Baseline, 4 weeks, 8 weeks and 12 weeks
  Amino acids, lipid metabolites, vitamins, neurotransmitters and other metabolites will be analyzed and tested using targeted metabolic analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Zhong Wang, Ph.D, Study Chair — China Academy of Chinese Science
Locations (1):
- Yuquan Hospital of Tsinghua University, Beijing, Beijing Municipality, China